CLINICAL TRIAL: NCT06696885
Title: Combined Effects of Mobile Based Video Games and Face to Face Exercise Program on Exercise Adherence and Hand Function in Chronic Stroke.
Brief Title: Mobile Applications for Exercise Adherence and Hand Function in Chronic Stroke.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0205
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Chronic Stroke Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A received mobile based video games along with task based training.
  Interventions: Other: Mobile based video games and task based training
- Group B (No Intervention): Group B received conventional physical therapy plan.

INTERVENTIONS:
Other: Mobile based video games and task based training — The experimental group received a mobile-based applications for 20 minutes and tasks-based training for 20 minutes per day (a total of 40 minutes), 6 days a week for 17 weeks. The time between each game was divided accordingly to work on improving hand function. The games and tasks were divided into three broad categories, Easy, Moderate, Difficult. Each category is applied for 6 weeks
  Arms: Group A

SUMMARY:
Stroke is a clinically defined syndrome characterized by an acute, focal neurological deficit due to vascular damage in the central nervous system. It is the second leading cause of death and disability globally. Stroke is not a singular disease but results from a variety of risk factors, disease processes, and mechanisms. Following a stroke, upper limb (UL) dysfunction affects 40-50% of individuals in the chronic phase, significantly impacting their ability to perform daily tasks. The latest trend in therapy involves the use of mobile video games within rehabilitation programs. These applications leverage the multi-touch interface of mobile devices to provide accurate monitoring of a patient's health status. Many of these mobile games are specifically designed to offer therapeutic tools that enhance dexterity and improve adherence to exercise routines.

DETAILED DESCRIPTION:
A Randomized Clinical Trail (RCT) design will be employed, conducted at Johar Pain Relief center over 10 months following the synopsis approval. The anticipated sample size, accounting for a 20% attrition rate will be 32 participants in each of the study groups. Group A will recieve mobile based video games along with task based therapy for exercise adherence and hand function while Group B will recieve conventional physical therapy. The sampling technique will be non probability convenience sampling with inclusion criteria of including chronic stroke patients aged between 30 to 75 years, both male and female genders are included in the study. The data collection tools include National Institute of Health Stroke Scale (NIHSS) , Fugl Meyer Assessment -UE (FM-UE) , Game User Experience Satisfaction Scale (GUESS) , Exercise Adherence Rating Scale (Ears) and Box and Block test was applied. The analysis will be conducted using SPSS for windows software version 25. Training session will last for 6 weeks which will be conducted 6 days a week. Mobile based video games and task based training will focus on exercise adherence and hand function, mainly focusing on hand dexterity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 30 to 75 years were included.
* Chronic stroke patients ranging from 6 months to 2 years (41).
* Participants having a stroke severity score > 6 on National Institute of Health Stroke Scale (NIHSS) (42).
* Modified Ashworth scale score ≤ 3 of the affected upper extremity (44).
* Montreal Cognitive Assessment (MoCA) score ≥ 26 (45).
* Patients who are able to sit without support.
* No contractures of the affected wrist and fingers.

Exclusion Criteria:

* Participants who show the symptoms of global or receptive aphasia.
* Participants who have medical problems or co-morbidities that interdict their participation in the study (such as shoulder pain in the paretic limb).
* Patients with severe apraxia, somatosensory problems.
* Severe spasticity of the affected wrist and finger flexors.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
• Fugl Meyer Assessment -UE (FM-UE) | 6 weeks
  FMA(UE) is a assessment tool for upper extremity which is divided into 5 domains (motor, sensory, balance, range of motion, and pain)
Game User Experience Satisfaction Scale (GUESS) | 6 weeks
  GUESS evaluates patient satisfaction of video-games following their participation in the gamified intervention. The GUESS consists of 55 items with 9 subscales. The subscales include usability/playability, narratives, play engrossment, enjoyment, creative freedom, audio aesthetics, personal gratification, social connectivity and visual aesthetics.
Exercise Adherence Rating Scale (EARS) | 6 weeks
  EARS is a tool designed to assess an individual's commitment to a prescribed exercise program.
Box and Block Test (BBT) | 6 weeks
  Box and Block Test (BBT) measures manual dexterity by counting how many blocks a participant can transfer between compartments in 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Binish Afzal, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sulfikar Ali A, Arumugam A, Kumaran D S. Effectiveness of an intensive, functional, gamified Rehabilitation program in improving upper limb motor function in people with stroke: A protocol of the EnteRtain randomized clinical trial. Contemp Clin Trials. 2021 Jun;105:106381. doi: 10.1016/j.cct.2021.106381. Epub 2021 Apr 20. PMID 33862286